CLINICAL TRIAL: NCT03151291
Title: Effects of Physical Exercise in the Form of Whole-body Electromyostimulation (WB-EMS) Combined With Individualized Nutritional Therapy Using Specific Dietary Supplements on Cancer Patients Undergoing Curative or Palliative Anti-cancer Treatment
Brief Title: Effects of WB-EMS and Specific Dietary Supplements on Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EMS and DS Tumor 01
Record Dates: First submitted 2017-05-11; First posted 2017-05-12 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Cancer; Cancer Cachexia; Weight Loss; Muscle Loss; Muscle Weakness
Keywords: cancer cachexia; WB-EMS; skeletal muscle mass; exercise; nutrition; dietary supplements
MeSH Terms: conditions — Neoplasms; Weight Loss; Muscular Atrophy; Muscle Weakness; Motor Activity | interventions — Carnitine; Eicosapentaenoic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Control group (No Intervention): "usual care" control group receives individualized nutritional support (dietary advices: daily protein intake > 1.0 g/kg bodyweight)
- EMS group (Experimental): physical exercise group performing a regular WB-EMS Training (two WB-EMS trainings per week; each session for 20 min)
  + individualized nutritional support (dietary advices: daily protein intake > 1.0 g/kg bodyweight)
  Interventions: Other: Whole-Body Electromyostimulation (WB-EMS)
- HMB group (Experimental): HMB supplemented group receives individualized nutritional support (dietary advices: daily protein intake > 1.0 g/kg bodyweight) + specific dietary supplementation with HMB (3 g/d)
  Interventions: Dietary Supplement: β-hydroxy-β-methylbutyrate (HMB)
- HMB+EMS group (Experimental): HMB supplemented physical exercise group performing a regular WB-EMS Training (two WB-EMS trainings per week; each session for 20 min)
  + individualized nutritional support (dietary advices: daily protein intake > 1.0 g/kg bodyweight) + specific dietary supplementation with HMB (3 g/d)
  Interventions: Dietary Supplement: β-hydroxy-β-methylbutyrate (HMB); Other: Whole-Body Electromyostimulation (WB-EMS)
- LC group (Experimental): LC supplemented group receives individualized nutritional support (dietary advices: daily protein intake > 1.0 g/kg bodyweight) + specific dietary supplementation with LC (4 g/d)
  Interventions: Dietary Supplement: L-carnitine (LC)
- LC+EMS group (Experimental): LC supplemented physical exercise group performing a regular WB-EMS Training (two WB-EMS trainings per week; each session for 20 min)
  + individualized nutritional support (dietary advices: daily protein intake > 1.0 g/kg bodyweight) + specific dietary supplementation with LC (4 g/d)
  Interventions: Dietary Supplement: L-carnitine (LC); Other: Whole-Body Electromyostimulation (WB-EMS)
- EPA group (Experimental): EPA supplemented group receives individualized nutritional support (dietary advices: daily protein intake > 1.0 g/kg bodyweight) + specific dietary supplementation with EPA (2.2 g/d)
  Interventions: Dietary Supplement: Eicosapentaenoic acid (EPA)
- EPA+EMS group (Experimental): EPA supplemented physical exercise group performing a regular WB-EMS Training (two WB-EMS trainings per week; each session for 20 min)
  + individualized nutritional support (dietary advices: daily protein intake > 1.0 g/kg bodyweight) + specific dietary supplementation with EPA (2.2 g/d)
  Interventions: Dietary Supplement: Eicosapentaenoic acid (EPA); Other: Whole-Body Electromyostimulation (WB-EMS)

INTERVENTIONS:
Dietary Supplement: β-hydroxy-β-methylbutyrate (HMB) — daily intake of 3 g HMB
  Arms: HMB group; HMB+EMS group
Dietary Supplement: L-carnitine (LC) — daily intake of 4 g LC
  Arms: LC group; LC+EMS group
Dietary Supplement: Eicosapentaenoic acid (EPA) — daily intake of 2.2 g EPA
  Arms: EPA group; EPA+EMS group
Other: Whole-Body Electromyostimulation (WB-EMS) — WB-EMS training is performed 2x/week for 12 weeks; Stimulation protocol: Frequency of 85 Hz, pulse duration of 0.35 ms, stimulation period of 6 sec, resting period of 4 sec; supervised by certified training instructors/physiotherapists participants perform simple exercises during the stimulation period following a video tutorial
  Arms: EMS group; EPA+EMS group; HMB+EMS group; LC+EMS group

SUMMARY:
Patients suffering from cancer often experience a loss of muscle mass and strength during disease and its therapy. Muscle wasting is the main characteristic of the so-called cancer cachexia syndrome and responsible for many therapy-related complications and a poorer prognosis of the patient. Stabilizing muscle mass should therefore be a great goal in cancer care. Physical exercise and nutrition are promising measures to combat cancer-related muscle atrophy but conventional exercise programs may not always be suitable for physical-weakened patients and increased catabolic processes are difficult to overcome by normal Nutrition - especially in advanced cancer. Therefore, the present study aims to test a combined approach of specific nutritional supplementation and exercise using the novel strength training method of Whole-Body electromyostimulation (WB-EMS). The study investigates the effect of a 12-week WB-EMS training combined with a dietary supplementation of β-hydroxy-β-methylbutyrate (HMB), L-carnitine (LC) or the omega-3-fatty acid eicosapentaenoic acid (EPA) on skeletal muscle mass, body composition, physical function, nutritional and inflammatory status, fatigue and quality of life in cancer patients undergoing oncological treatment. The results of this study may help to clarify the effectiveness of those combined interventions to counteract muscle wasting and other symptoms of cancer cachexia.

ELIGIBILITY:
Inclusion Criteria:

* malignant disease (solid or hematological cancer) e.g. head and neck cancer, colorectal carcinoma, small intestinal cancer, gastric cancer, oesophageal cancer, pancreas carcinoma, liver cell carcinoma, cholangiocarcinoma,lung cancer, breast cancer, cervix cancer, ovarian cancer, prostate cancer, renal cell carcinoma, malignant melanoma, patients with leukaemia and malignant lymphomas
* ECOG Performance Status ≤ 2

Exclusion Criteria:

* simultaneous participation in other nutritional or exercise intervention trials
* acute cardiovascular events
* use of anabolic medications
* epilepsy
* severe neurological diseases
* skin lesions in the area of electrodes
* energy active metals in body
* pregnancy
* acute vein thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Skeletal muscle mass | 12 weeks
  Skeletal muscle mass assessed by bioelectrical impedance analysis (in kg)

SECONDARY OUTCOMES:
Physical function - isometric muscle strength | 12 weeks
  Isometric hand grip strength assessed by hand Dynamometer (in kg)
Physical function - Endurance | 12 weeks
  Six-minute-walk test (walking distance in m)
Physical function - Lower limb strength | 12 weeks
  30 second sit-to-stand test (number of sit-to-stand cycles)
Patient-reported performance status | 12 weeks
  ECOG performance status/Karnofsky index
Patient-reported Quality of Life (QoL) | 12 weeks
  EORTC QLQ - C30 questionnaire
Patient-reported Fatigue | 12 weeks
  FACIT-Fatigue scale
Inflammatory blood markers | 12 weeks
  Blood collection and analysis of e.g. C-reactive protein (CRP), Albumin

CONTACTS AND LOCATIONS:
Locations (1):
- Hector-Center for Nutrition, Exercise and Sports, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No